CLINICAL TRIAL: NCT05360277
Title: Maintenance Tislelizumab Combined With Capecitabine to Treat Metastatic Colorectal Cancer With No Evidence of Disease
Brief Title: Maintenance Tislelizumab + Capecitabine to Treat Metastatic Colorectal Cancer
Acronym: CAMCO2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Professer, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG-C02; GIHSYSU-24 (Other: The Sixth Affiliated Hospital of Sun Yat-sen University)
Record Dates: First submitted 2022-04-30; First posted 2022-05-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Colorectal Cancer，NED
Keywords: Metastatic Colorectal Cancer，NED
MeSH Terms: interventions — tislelizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + Capecitabine (Experimental): Tislelizumab 200mg every 3 weeks, or 1 year after completion of perioperative chemotherapy.
  Capecitabine was given at a dose of 850 mg/m2 twice a day by mouth, 2 weeks on/ 1 week off, for 1 year after completion of perioperative chemotherapy.
  Interventions: Drug: Tislelizumab + Capecitabine
- Best supportive care (Active Comparator): Best supportive care was the standard care in this setting.
  Interventions: Other: Best supportive care

INTERVENTIONS:
Drug: Tislelizumab + Capecitabine — Tislelizumab 200mg iv every 3 weeks, for 1 year after completion of perioperative chemotherapy.
  Capecitabine was given at a dose of 850 mg/m2 twice a day by mouth, 2 weeks on/ 1 week off, for 1 year after completion of perioperative chemotherapy.
  Arms: Tislelizumab + Capecitabine
Other: Best supportive care — Best supportive care
  Arms: Best supportive care

SUMMARY:
Surgery with integrated treatment for metastatic colorectal cancer (mCRC) has created a new clinical setting known as mCRC with no evidence of disease (NED). However, these patients have a high risk of developing persistent cancer. This study aimed to investigate the efficacy and safety of Tislelizumab combined with capecitabine as a maintenance treatment for patients with mCRC-NED.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, open-label, single-center study designed to compare the efficacy and safety of tislelizumab+ capecitabine versus best-supported care as a first-line maintenance treatment in participants with mCRC-NED.

Patients who underwent synchronously or staged removal of primary and metastatic lesions, achieving NED, and histologically confirmed colorectal adenocarcinoma were recruited in this trial. The primary endpoint was disease-free survival (DFS). Secondary endpoints included overall survival (OS) and adverse events. This study will provide novel data on the efficacy and safety profile of the combination of tislelizumab and capecitabine in patients with mCRC-NED.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years, < 80 years
2. Written informed consent
3. Histologically or cytologically confirmed CRC
4. Surgery with integrated treatment for metastatic colorectal cancer (mCRC) and achieved a statute of no evidence of disease (NED), as determined by a multidisciplinary tumor board.
5. cytoreduction surgery achieves CC0 (no visible residual tumor) if there is peritoneal metastasis
6. No previous chemotherapy
7. Synchronous or metachronous metastatic disease: maximum of two distant organs or regions involved
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
9. Adequate hematologic and organ function

Exclusion Criteria:

1. Presence of any other active cancer
2. Presence of active infections requiring antibiotics
3. History of active autoimmune disease requiring systemic treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 36 months
  The time from NED to the first occurrence of any of the following events: local relapse, distant metastasis, or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 60 months
  The time from NED to death from any cause
Adverse events | 60 months
  Side effect of both agents

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No